# Official Title: Effect of Emotion Mindsets on Emotion Processing: A Multilevel Experimental Investigation

NCT Number: 03978871

Date of final version of consent: July 29th, 2020

# UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN



#### ADOLESCENT ASSENT FORM

**Title of study:** Study of Teen Emotion Processing (STEP)

Principal Investigator/s: Dr. Karen Rudolph, Dr. Wendy Heller, & Dr. Sepideh Sadaghiani

Contact information is listed on p. 3.

**Department/s:** Psychology, University of Illinois at Urbana-Champaign

#### Research project:

The purpose of this research is to examine emotion processing in adolescents and to help individuals develop adaptive ways of dealing with their emotions. The study involves completing questionnaires, viewing video clips, and participating in a debriefing discussion with a staff member. Study participation will take approximately 150 minutes.

#### **Procedures:**

- 1) You will be asked to fill out a number of questionnaires. The types of topics addressed in the questionnaires include emotions, behaviors, and experiences, including questions specific to your experiences during the COVID-19 pandemic. Example questions include "I felt unhappy or miserable," "I cheer up quickly," and "How many people close to you were diagnosed with COVID." These questions should take no more than 30 minutes to complete. The questionnaires can be completed using a secure on-line website or on paper.
- 2) You will be asked to participate in a role play where you will talk about friendships. There will be parts of your visit that are recorded but we will not share any answers or recordings without your permission. While the completion of this task has the potential to cause mild discomfort, it is expected to be similar to any act of public speaking.
- 3) You will be asked to view brief video clips and rate how you feel after viewing them. Some of the video clips you will view are moderately negative. While viewing these video clips may cause mild discomfort, they do not pose any risk. The images you view may cause mild discomfort because they may remind you of negative experiences in your own life. If you report higher than baseline ratings on a measure of your emotions at the end of the study, we will follow-up with you the following day.
- 4) You will complete a computer task in which you push a button whenever you see a letter except the letter "x."
- 5) You will be asked to complete a computer-administered session in which you will learn about adolescent development and some basic information about the brain. We will also ask you to

#### A2. Adolescent Assent

provide information to younger adolescents based on what you learned. This computer session will last approximately 30 minutes.

6) Finally, project staff will conduct a debriefing session with you. The purpose of this session is for our staff to ask questions and receive feedback from participants on certain measures and aspects of our study. For example, project staff may ask if any words or items were confusing to you. Project staff may take hand-written notes of your responses during this part.

All procedures will be employed with sensitivity to your feelings. To avoid any discomfort, you may skip questions you do not want to answer. Your participation in this study is voluntary, and you may withdraw from the study at any time without penalty.

You will be offered breaks periodically throughout the study session. You are encouraged to notify the researchers that you need to take a break at any time. Restrooms and drinking water will be available during study sessions.

#### **Remuneration:**

You will receive \$50 for your participation. If your participation is discontinued (by you, your parent, or the experimenter), you will be paid according to your level of participation.

#### **Risks & Benefits:**

You will be asked to report on sensitive topics, including your emotions. While these questions are sensitive in nature, answering them does not pose any expected risk to you. Your responses will be completely confidential and voluntary and you may choose not to respond to any questions that you are uncomfortable with. The answers to your questions will not be shared with anyone except our research team unless we are concerned about you or someone else's safety.

There is no direct personal benefit to participating in this study. However, your participation provides the investigator with a greater understanding about emotional development in youth. The study results may be used to help other people in the future.

### **Confidentiality:**

All possible steps have been taken to assure your privacy. The experimenter will assign you an arbitrary code number which will be used throughout the study. Only this code (and never your name) will be used when analyzing or reporting the data. Any identifying information will be kept in a locked location in the Investigator's laboratory. In addition, laws and University rules might require that the research data be made available to the following groups: 1) representatives of the University committee and office that reviews and approves research studies, such as the Institutional Review Board (IRB) or Office for Protection of Research Subjects; 2) representatives of the state and University responsible for ethical, regulatory, or financial oversight of research; and, 3) research collaborators at the Biomedical Imaging Center. Anyone who accesses the research data will be required to maintain the confidentiality of any and all participants.

# Voluntary participation and withdrawal:

Participation in the research is voluntary. You are free to stop participating at any time. If you choose not to volunteer, or if the research is ended for any reason by you, your parent, or the researchers, it will have no effect on any other benefits to which you are entitled. If you are a student at the University of Illinois, your decision to participate, decline, or withdraw from participation will have no effect on your grades at, status at, or future relationships with the university.

## **Dissemination of findings:**

The results of the research may be published and presented at lectures and professional meetings, but you will not be identified in any such publication or presentation.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify your child. At most, the Web site will include a summary of the results of the research project. You can search this website at any time.

#### **Contact Information:**

You will be given a copy of this consent form for your records. If at any time, either now or later, you have a question, please feel free to ask it. If you have questions or concerns regarding your rights as a participant in this study, please contact the University of Illinois Institutional Review Board office at (217) 333-2670 or <a href="mailto:irb@illinois.edu">irb@illinois.edu</a>. If you have any questions about this particular study, you may contact Dr. Karen Rudolph at (217)333-8624 or <a href="mailto:krudolph@illinois.edu">krudolph@illinois.edu</a>, Dr. Wendy Heller at (217)244-8249 or <a href="mailto:krudolph@illinois.edu">w-heller@illinois.edu</a>, or Dr. Sepideh Sadaghiani at (217)300-2566 or <a href="mailto:sepideh@illinois.edu">sepideh@illinois.edu</a>.

If you feel you have not been treated according to the descriptions in this form, or if you have any questions about your rights as a research subject, including questions, concerns, complaints, or to offer input, you may call the Office for the Protection of Research Subjects (OPRS) at 217-333-2670 or e-mail OPRS at irb@illinois.edu.

#### **Agreement:**

By signing this document, I am stating that the nature of the study has been explained to me. I am also stating that I have had the opportunity to ask questions concerning any and all aspects of the procedures involved. I am also aware that participation is voluntary, that I may withdraw my consent at any time, and that if I decide not to participate or decide to withdraw participation, I will not be penalized in any way.

| Name: | |
|------------|------|
| Signature: | <br> |
| Date: | |

I, the undersigned, hereby consent to be a participant in the project described above.